CLINICAL TRIAL: NCT04513262
Title: Effects of Pneumoperitoneum on Ventilatory Parameters in Patients Undergoing Video-assisted Surgery
Brief Title: Effects of Video-Assisted Surgery on Ventilatory Parameters
Status: Completed | Type: Observational
Sponsor: Institutul Clinic Fundeni (Other)
Responsible Party: Principal Investigator, Popescu Mihai, Clinical Professor, Institutul Clinic Fundeni
Other Study IDs: RAS
Record Dates: First submitted 2020-08-11; First posted 2020-08-14 (Actual); Last update posted 2020-08-14 (Actual); Status verified 2020-08

CONDITIONS: Surgery--Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Video-assisted surgery: Patients undergoing video-assisted major abdominal surgery (VAS) in Trendelenburg position. The decision regarding the type of VAS was made by the attending surgeon prior to study inclusion. Twenty-five consecutive patients undergoing classic laparoscopic surgery and twenty-five patients undergoing robotic-assisted surgery will be included in the study.
  Interventions: Procedure: mechanical ventilation during video-assisted surgery

INTERVENTIONS:
Procedure: mechanical ventilation during video-assisted surgery — observed variation of ventilatory parameters during video-assisted surgery

SUMMARY:
The study investigates the effects of induced pneumoperitoneum during surgery on ventilatory parameters including peak inspiratory pressure, lung compliance, end-tidal CO2 at specific time-points: after induction of anaesthesia, after induction of surgery, one-hour and two-hours during surgery, end of surgery.

The effects of pneumoperitoneum are compared between two groups of patients: patients undergoing laparoscopic surgery and patients undergoing robotic-assisted surgery. No intervention was performed in this study and the decision for type of surgery performed was made by the attending surgeon prior to study inclusion

ELIGIBILITY:
Inclusion Criteria:

* patients who underwent video-assisted surgery by either classic laparoscopy or robotic-assisted surgery.

Exclusion Criteria:

* refusal to participate
* conversion of surgery to laparotomy
* need of vasopressure support
* preoperative severe respiratory dysfunction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: consecutive patients undergoing video-assisted surgery in a university hospital after inclusion and exclusion criteria have been met. Video-assisted surgery is defined by either classic laparoscopic surgery or robotic assisted surgery and the medical decision between the two types of surgery was performed by the attending surgeon prior to patient inclusion (unrelated to the study).
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2015-03-20 (Actual); Primary Completion 2018-11-10 (Actual); Study Completion 2018-11-10 (Actual)

PRIMARY OUTCOMES:
lung compliance | one-hour and two-hours after induction of pneumoperitoneum
  change in lung compliance (mL/cmH2O) before and after induction of pneumoperitoneum in patients undergoing VAS. Lung compliance is automatically calculated by the anesthesia machine during surgery. The study compares the magnitude in change associated with VAS.

SECONDARY OUTCOMES:
arterial to end-tidal CO2 difference | one-hour and two-hours after induction of pneumoperitoneum
  difference in arterial to end-tidal CO2 (mmHg) during surgery. Arterial blood samples and end-tidal CO2 were simultanously obtained at the specific time-points.

CONTACTS AND LOCATIONS:
Overall Officials: Dana Tomescu, Prof, Study Chair — Fundeni Clinical Institute
Locations (1):
- Fundeni Clinical Institute, Bucharest, Romania

IPD SHARING:
Plan to Share IPD: No